CLINICAL TRIAL: NCT03805295
Title: Implementation and Evaluation of a Before School Physical Activity Program in Revere, MA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Council on Exercise (Other); BOKS (Unknown)
Responsible Party: Principal Investigator, Elsie Taveras, MD, Chief, Division of General Pediatrics, Massachusetts General Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2017P002770
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Overweight and Obesity; Physical Activity; Quality of Life; Fitness; Executive Function
MeSH Terms: conditions — Overweight; Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spring 2018 Participation (Experimental): Students in this arm (40 per school, up to 120 total) will participate in the BOKS program in Winter-Spring 2018. They will serve as the control group in Fall 2018.
  Interventions: Other: BOKS Program
- Fall 2018 Participation (Experimental): Students in this arm (40 per school, up to 120 total) will participate in the BOKS program in Fall 2018.
  Interventions: Other: BOKS Program

INTERVENTIONS:
Other: BOKS Program — 12-week physical activity program, occurring 3x/week, lasting 30-60 minutes per session.

SUMMARY:
This study evaluates the implementation of the BOKS program in three schools (K-8) in Revere, MA, and its effect on participating students with regard to BMI, cognitive, and quality of life outcomes. BOKS (Build Our Kids' Success) is a before-school physical activity program that has been implemented in over 2,000 elementary and middle schools. Two sessions will be held (Spring 2018 and Winter 2018. This is a cohort study evaluating the impact of program participation on child BMI, quality of life, and executive function.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the BOKS program
* Participating school
* Age 5-14

Exclusion Criteria:

* No valid consent
* Not enrolled in BOKS

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 188 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elsie Taveras, MD, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Spring 2018 Participation | Fall 2018 Participation
Started | 103 | 85
Completed | 86 | 42
Not Completed | 17 | 43
Not completed — Lost to Follow-up | 17 | 43

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Spring 2018 Participation | Fall 2018 Participation | Total
Number analyzed (Participants) | 86 | 42 | 128
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 86 | 42 | 128
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.2 (2.2) | 9.2 (2.2) | 9.2 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 26 | 67
  Male | 45 | 16 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 21 | 52
  Not Hispanic or Latino | 43 | 14 | 57
  Unknown or Not Reported | 12 | 7 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 2 | 8
  White | 51 | 30 | 81
  More than one race | 13 | 2 | 15
  Unknown or Not Reported | 12 | 7 | 19
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 86 | 42 | 128

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Mass Index (kg/m^2)
Description: calculated from height and weight
Time Frame: Baseline, Follow-up for each session (12 weeks)
Measure: Mean (Standard Deviation); unit: kg/m^2 (BMI change)
Arm/Group | Spring 2018 Participation | Fall 2018 Participation
Number analyzed (Participants) | 76 | 31
kg/m^2 (BMI change) | 0.14 (0.63) | 0.01 (0.70)

2. Secondary Outcome: Change in Executive Function
Description: Executive function and attention/concentration as measured by the Flanker Task
Time Frame: Baseline, Follow-up for each session (12 weeks)
Reporting Status: Not Posted

3. Secondary Outcome: Change in Quality of Life PedsQL
Description: Measured by PedsQL, a validated measure of pediatric self-rated quality of life with higher score indicating higher quality of life.
Time Frame: Baseline, Follow-up for each session (12 weeks)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Spring 2018 Participation | Fall 2018 Participation
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/42
Other Adverse Events (participants affected / at risk) | 0/86 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-09): https://cdn.clinicaltrials.gov/large-docs/95/NCT03805295/Prot_SAP_000.pdf
  • Informed Consent Form (2018-08-14): https://cdn.clinicaltrials.gov/large-docs/95/NCT03805295/ICF_001.pdf